CLINICAL TRIAL: NCT02204982
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of Duvelisib in Combination With Rituximab vs Rituximab in Subjects With Previously Treated Follicular Lymphoma
Brief Title: Study of Duvelisib in Combination With Rituximab vs Rituximab in Subjects With Previously Treated Follicular Lymphoma
Acronym: DYNAMO + R
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor is focusing on studies which can enable registration of duvelisib
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPI-145-08; 2013-002406-31 (EudraCT Number)
Record Dates: First submitted 2014-07-25; First posted 2014-07-31 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Follicular Lymphoma
Keywords: Phase 3, Follicular Lymphoma, FL, PI3K
MeSH Terms: conditions — Lymphoma, Follicular; Hereditary Sensory and Autonomic Neuropathies | interventions — duvelisib; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duvelisib + Rituximab (Experimental): Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules.
  Rituximab is administered as an intravenous (IV) infusion and is supplied in single-use vials at two strengths, 100 mg and 500 mg.
  Interventions: Drug: Duvelisib; Drug: Rituximab
- Placebo + Rituximab (Placebo Comparator): Placebo is administered orally and supplied as formulated capsules to match the active 5 mg and 25 mg capsules.
  Rituximab is administered as an intravenous (IV) infusion and is supplied in single-use vials at two strengths, 100 mg and 500 mg.
  Interventions: Drug: Placebo; Drug: Rituximab

INTERVENTIONS:
Drug: Duvelisib — PI3K Inhibitor
  Other Names: Copiktra, IPI-145
  Arms: Duvelisib + Rituximab
Drug: Placebo — Matching Placebo (25 mg BID) administered orally in 28-day continuous treatment cycles.
  Arms: Placebo + Rituximab
Drug: Rituximab — IV infusion of rituximab (375 mg/m2) once weekly for 4 weeks during Cycle 1, then once on Day 1 of Cycles 4, 6, 8, and 10.
  Other Names: Rituxan; MabThera

SUMMARY:
A study to evaluate the safety and efficacy of duvelisib administered in combination with rituximab vs placebo in combination with rituximab in patients with previously treated CD20-positive follicular lymphoma who are not suitable candidates for chemotherapy.

DETAILED DESCRIPTION:
Study IPI-145-08 is an international, multicenter, randomized, double-blind, placebo-controlled, parallel-group, Phase 3 study designed to evaluate the efficacy and safety of duvelisib in combination with rituximab vs placebo in combination with rituximab in subjects with previously treated CD20-positive follicular lymphoma.

Approximately 400 subjects will receive 25 mg of duvelisib or placebo, orally BID for 28 day continuous cycles, in combination with 375 mg/m2 of Rituximab given once weekly for 4 weeks during Cycle 1 and then once on Day 1 of Cycles 4, 6, 8, and 10. Patients will remain on treatment for up to 27 cycles and may continue treatment if clinical benefit is observed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20-positive FL:

  * Histology grades 1, 2 or 3a
  * Biopsy-confirmed histopathological diagnosis of FL. Biopsy specimen should be obtained ≤2 years prior to randomization, unless medically contraindicated
* CD20 immunophenotyping performed ≤2 years prior to randomization
* First or subsequent relapse following at least one induction therapy regimen containing rituximab in combination with an anthracycline or rituximab in combination with an alkylating agent
* Patients in first relapse must be chemoresistant or intolerant to chemotherapy
* No response or disease progression ≤ 24 months from start of last previous therapy
* At least 1 measurable disease lesion >1.5 cm in at least one diameter by CT/CT-PET or magnetic resonance imaging (MRI) in an area of no prior radiation therapy, or in an area that was previously irradiated that has documented progression

Exclusion Criteria:

* Clinical evidence of other indolent forms of lymphoma (e.g., marginal zone lymphoma [MZL], small lymphocytic lymphoma [SLL])
* Transformation to a more aggressive subtype of lymphoma or grade 3b FL
* Refractory to rituximab: defined as disease progression while receiving or within 6 months of completing either weekly rituximab induction therapy, or rituximab-based chemoimmunotherapy induction
* Intolerance to rituximab or severe allergic or anaphylactic reaction to any humanized or murine monoclonal antibodies
* Prior allogeneic hematopoietic stem cell transplant (HSCT)
* Known Central Nervous System (CNS) lymphoma; subjects with symptoms of CNS disease must have a negative CT scan and negative diagnostic lumbar puncture
* Prior treatment with a PI3K inhibitor or BTK inhibitor
* History of tuberculosis within the preceding two years
* Ongoing systemic bacterial, fungal, or viral infections at randomization (defined as requiring IV antimicrobial, antifungal or antiviral agents)
* Subjects on antimicrobial, antifungal or antiviral prophylaxis are not specifically excluded if all other I/E criteria are met
* Prior, current, or chronic hepatitis B or hepatitis C infection, positive result for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) or hepatitis C virus antibodies (HCV Ab)
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Youssoufian, MD, Study Chair — Verastem, Inc.
Locations (5):
- Frankston, Victoria, Australia
- Bordeaux, France
- Italy (2):
  - Bologna
  - Terni
- Gdynia, Poland

RESULTS

PARTICIPANT FLOW:
Groups:
- Duvelisib + Rituximab: Duvelisib is administered orally and supplied as 5 mg and 25 mg formulated capsules.
  Rituximab is administered as an intravenous (IV) infusion and is supplied in single-use vials at two strengths, 100 mg and 500 mg.
  Duvelisib: duvelisib (25 mg BID) administered orally in 28-day continuous treatment cycles
  Rituximab: IV infusion of rituximab (375 mg/m2) once weekly for 4 weeks during Cycle 1, then once on Day 1 of Cycles 4, 6, 8, and 10.
- Placebo + Rituximab: Placebo is administered orally and supplied as formulated capsules to match the active 5 mg and 25 mg capsules.
  Rituximab is administered as an intravenous (IV) infusion and is supplied in single-use vials at two strengths, 100 mg and 500 mg.
  Placebo: Matching Placebo (25 mg BID) administered orally in 28-day continuous treatment cycles.
  Rituximab: IV infusion of rituximab (375 mg/m2) once weekly for 4 weeks during Cycle 1, then once on Day 1 of Cycles 4, 6, 8, and 10.
Period: Overall Study
Arm/Group | Duvelisib + Rituximab | Placebo + Rituximab
Started | 6 | 7
Completed | 2 | 0
Not Completed | 4 | 7
Not completed — Patient ineligible-medical monitor | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Adverse Event and Investigator decision | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Protocol-Specified Disease Progression | 0 | 4
Not completed — Termination of Study bySponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duvelisib + Rituximab | Placebo + Rituximab | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 2 | 5 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.5 [55 to 77] | 68 [47 to 79] | 68 [55 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 2 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 5 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 2
  Australia | 1 | 0 | 1
  Italy | 2 | 1 | 3
  Spain | 1 | 1 | 2
  Poland | 1 | 2 | 3
  Canada | 0 | 1 | 1
  France | 0 | 1 | 1
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants]
  0=Fully active, no restrictions | 4 | 6 | 10
  1= Restricted in physically strenuous activity | 2 | 1 | 3
  2=Ambulatory more than 50% of waking hours | 0 | 0 | 0
  3=Confined to bed or chair more than 50% of waking | 0 | 0 | 0
  4=Completely disabled | 0 | 0 | 0
  5=Dead | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Due to the small number of enrolled subjects and study being terminated, PFS endpoint analysis was not performed.
Time Frame: Until disease progression, for up to 5 years from randomization
Population: Data could not be reported because the study was terminated early and a sufficient number of subjects and events were not available for analysis.
Arm/Group | Duvelisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Response Rate (ORR)
Time Frame: Until disease progression, for up to 5 years from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Duvelisib + Rituximab | Placebo + Rituximab
Number analyzed (Participants) | 5 | 6
Participants
  Complete Response | 3 | 0
  Partial Response | 2 | 1
  Stable Disease | 0 | 3
  Progressive Disease | 0 | 2

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Duvelisib + Rituximab | Placebo + Rituximab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 5/6 | 0/7
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib + Rituximab (N=6) | Placebo + Rituximab (N=7)
Pneumonia (Infections and infestations) | 2 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 0
Chronic Obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Duvelisib + Rituximab (N=6) | Placebo + Rituximab (N=7)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Amylase increased (Investigations) | 1 | 0
Blood Cholesterol increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Blood Uric acid increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 2 | 2
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 1
Chills (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Influenza like illness (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes